CLINICAL TRIAL: NCT02565706
Title: Online WIC Nutrition Education to Promote Farmers' Market Fruit and Vegetable Purchases and Consumption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: William Paterson University of New Jersey (Other)
Collaborators: USDA Food and Nutrition Service (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jennifer Di Noia, Professor, William Paterson University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WIC NEI-12-TX
Record Dates: First submitted 2015-09-29; First posted 2015-10-01 (Estimated); Results first posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Cardiovascular Diseases; Cancer; Type 2 Diabetes; Obesity
Keywords: Fruit, vegetables, income, WIC program, farmers' market
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- WIC Fresh Start Program (Active Comparator): Participants in this arm receive the Fresh Start program.
  Interventions: Behavioral: WIC Fresh Start Program
- Existing Online Health Education (Active Comparator): Participants in this arm receive existing online WIC health education.
  Interventions: Behavioral: Existing Online Health Education
- WIC Fresh Start Program (FMNP) (Experimental): Participants in this arm receive the Fresh Start program and WIC Farmers' Market Nutrition Program (FMNP) vouchers redeemable at farmers' markets.
  Interventions: Behavioral: WIC Fresh Start Program
- Existing Online Health Education (FMNP) (Active Comparator): Participants in this arm receive existing online WIC health education and WIC Farmers' Market Nutrition Program (FMNP) vouchers redeemable at farmers' markets.
  Interventions: Behavioral: Existing Online Health Education

INTERVENTIONS:
Behavioral: WIC Fresh Start Program — The intervention is an online lesson to promote farmers' market FV purchases and consumption. The lesson comprises three modules, each consisting of 1) behavior change content presented through a video segment featuring WIC participants, and 2) an interactive activity to build targeted knowledge, attitudes, and skills.
  Arms: WIC Fresh Start Program; WIC Fresh Start Program (FMNP)
Behavioral: Existing Online Health Education — Any of seven existing online WIC health education lessons (lessons are available on breastfeeding, being active, fruits and vegetables, calcium, cholesterol, oral health and iron). The lessons consist of an introductory segment presented with online text and graphics. After reading this material, viewers have the option to complete one of four lesson activities. The activities provide opportunities for viewers to read further on the topic and are designed to reinforce key points of the lesson.
  Arms: Existing Online Health Education; Existing Online Health Education (FMNP)

SUMMARY:
This study is evaluating the WIC Fresh Start program, a theory-driven, web-based nutrition education lesson to promote farmers' market fruit and vegetable purchases and consumption among women enrolled in the Special Supplemental Nutrition Program for Women, Infants and Children (WIC).

DETAILED DESCRIPTION:
This study is evaluating the WIC Fresh Start program, a theory-driven, web-based nutrition education lesson to promote fruit and vegetable (FV) consumption among women enrolled in the Special Supplemental Nutrition Program for Women, Infants and Children (WIC). Designed to leverage vouchers provided to WIC participants for FV purchases through the Farmers' Market Nutrition Program (FMNP) and monthly cash value vouchers (CVVs) redeemable at farmers' markets, the lesson is conceptually grounded in formative research on knowledge, attitudes and skills influencing farmers' market FV purchases and consumption and theoretical understanding of approaches for modifying them. Lesson content delivery is primarily through short video segments and audio output to increase accessibility for low-literate learners. Informed by a community-based participatory research approach, WIC participants are engaged as full partners in the development of the lesson and the delivery of content (videos feature WIC participants). The setting is a large WIC agency serving three New Jersey counties. Separate samples of women were recruited to participate in 1) focus groups for guiding lesson content development (N = 56 participants) and pretesting the resulting content (N = 52 participants), 2) cognitive testing to assess the clarity and interpretability of items and response formats in measures of knowledge, attitudes and skills developed for the study (N = 15), 3) one-on-one sessions to assess reactions to initial versions of video segments developed for the lesson (N = 20), and 4) the outcome evaluation (N = 744). Stratified based on FMNP voucher receipt, participants are randomized to receive the lesson or existing online health education. Outcome measures (administered orally to reduce literacy demands of the response task) are completed at pretest (immediately before the lesson), posttest (two weeks after the lesson), and 3 and 6 months after posttesting. Short- and long-term lesson effects on FV intake, FMNP voucher redemption and the redemption of CVVs at farmers' markets will be evaluated. Evidence for mediation by knowledge, attitudes, and skills of lesson effects on FV intake and voucher redemption, dose-response relationships, and user satisfaction with the lesson also will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant or postpartum WIC participant
* Female caregiver of infant/child WIC participant

Exclusion Criteria:

* Restrictions on food intake
* Classified by WIC as high risk/requiring an individualized nutrition care plan

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 744 (Actual)
Dates: Start 2014-07; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Di Noia, PhD, Principal Investigator — Professor, Department of Sociology, William Paterson University
Locations (1):
- Saint Joseph's WIC Program, Paterson, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
The data sets used and/or analyzed during this study are available from the corresponding author on reasonable request.
Time Frame: Data are available for sharing.
Access Criteria: Contact the PI with requests (dinoiaj@wpunj.edu).

REFERENCES:
- [Background] Di Noia J, Monica D, Sikorskii A, Cullen KW. Outcomes of a randomized controlled trial of nutrition education to promote farmers' market fruit and vegetable purchases and consumption among women enrolled in the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC). BMC Nutr. 2017 Jun 21;3:48. doi: 10.1186/s40795-017-0172-0. eCollection 2017. PMID 32153828
- [Background] Di Noia J, Monica D, Cullen KW, Perez-Escamilla R, Gray HL, Sikorskii A. Differences in Fruit and Vegetable Intake by Race/Ethnicity and by Hispanic Origin and Nativity Among Women in the Special Supplemental Nutrition Program for Women, Infants, and Children, 2015. Prev Chronic Dis. 2016 Aug 25;13:E115. doi: 10.5888/pcd13.160130. PMID 27560723
- [Background] Di Noia J, Cullen KW, Monica D. Social Desirability Trait Is Associated with Self-Reported Vegetable Intake among Women Enrolled in the Special Supplemental Nutrition Program for Women, Infants, and Children. J Acad Nutr Diet. 2016 Dec;116(12):1942-1950. doi: 10.1016/j.jand.2016.07.008. Epub 2016 Sep 21. PMID 27665255
- [Background] Di Noia J, Monica D, Cullen KW, Thompson D. Perceived Influences on Farmers' Market Use among Urban, WIC-enrolled Women. Am J Health Behav. 2017 Sep 1;41(5):618-629. doi: 10.5993/AJHB.41.5.11. PMID 28760184
- [Result] Di Noia J, Monica D, Gray HL, Cullen KW. The Special Supplemental Nutrition Program for Women, Infants, and Children Fresh Start Randomized Controlled Trial: Baseline Participant Characteristics and Reliability of Measures. J Acad Nutr Diet. 2016 Dec;116(12):1899-1913. doi: 10.1016/j.jand.2016.07.020. Epub 2016 Sep 20. PMID 27663256

RESULTS

PARTICIPANT FLOW:
Groups:
- WIC Fresh Start Program: Participants in this arm receive the Fresh Start program.
  The Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) Fresh Start Program: The intervention is an online lesson to promote farmers' market fruit and vegetable (FV) purchases and consumption. The lesson comprises three modules, each consisting of 1) behavior change content presented through a video segment featuring WIC participants, and 2) an interactive activity to build targeted knowledge, attitudes, and skills.
Period: Overall Study
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Started | 178 | 172 | 193 | 201
Completed | 101 | 90 | 104 | 116
Not Completed | 77 | 82 | 89 | 85
Not completed — Withdrawal by Subject | 5 | 7 | 7 | 11
Not completed — Lost to Follow-up | 72 | 75 | 82 | 74

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP) | Total
Number analyzed (Participants) | 178 | 172 | 193 | 201 | 744
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.83 (7.31) | 28.89 (6.56) | 29.25 (6.44) | 28.91 (7.03) | 28.97 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 178 | 172 | 193 | 201 | 744
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American | 59 | 47 | 47 | 68 | 221
  Hispanic | 103 | 99 | 124 | 110 | 436
  White or other | 9 | 22 | 17 | 18 | 66
  Two or more races | 4 | 3 | 3 | 4 | 14
  Missing | 3 | 1 | 2 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 178 | 172 | 193 | 201 | 744

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Redeemed FMNP Vouchers
Description: The state WIC agency is providing data on FMNP voucher redemption.
Time Frame: 6 months (2015 farmers' market season [June to November 2015])
Measure: Number; unit: participants
Arm/Group | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 193 | 201
participants | 84 | 77

2. Primary Outcome: Frequency of Fruit and Vegetable Intake
Description: Times per day fruits and vegetable are consumed as assessed by a validated food frequency questionnaire.
Time Frame: Pretest, posttest (2 weeks after pretest), and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Times per day consumed
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Times per day consumed
  Posttest | 3.71 (.18) | 4.00 (.18) | 3.88 (.16) | 3.90 (.17)
  3-month follow-up | 3.85 (.19) | 3.44 (.20) | 3.70 (.18) | 3.51 (.17)
  6-month follow-up | 3.90 (.22) | 3.78 (.23) | 3.41 (.21) | 3.26 (.20)

3. Primary Outcome: Quantity of Fruit and Vegetable Intake
Description: Cups per day consumed of fruits and vegetables as assessed by a validated fruit and vegetable screener.
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Population: Data are reported for the 6-month follow-up assessment.
Measure: Least Squares Mean (Standard Error); unit: Cups per day consumed
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Cups per day consumed
  Posttest | 4.49 (.21) | 4.61 (.21) | 4.54 (.19) | 4.44 (.19)
  3-month follow-up | 4.87 (.23) | 4.67 (.23) | 4.93 (.21) | 4.75 (.20)
  6-month follow-up | 4.74 (.26) | 4.91 (.27) | 4.76 (.24) | 4.88 (.23)

4. Secondary Outcome: Number of Participants Who Redeemed Cash Value Vouchers at Farmers' Markets
Description: The state WIC agency is providing data on cash value voucher redemption.
Time Frame: 6 months (2015 farmers' market season [June to November 2015])
Measure: Count of Participants; unit: Participants
Groups:
- WIC Fresh Start Program (FMNP): Participants in this arm receive the Fresh Start program (includes those who receive WIC Farmers' Market Nutrition Program [FMNP] vouchers and those who do not).
  WIC Fresh Start Program: The intervention is an online lesson to promote farmers' market FV purchases and consumption. The lesson comprises three modules, each consisting of 1) behavior change content presented through a video segment featuring WIC participants, and 2) an interactive activity to build targeted knowledge, attitudes, and skills.
- Existing Online Health Education (FMNP): Participants in this arm receive existing online WIC health education (includes those who receive WIC Farmers' Market Nutrition Program [FMNP] vouchers and those who do not).
  Existing Online Health Education: Any of seven existing online WIC health education lessons (lessons are available on breastfeeding, being active, fruits and vegetables, calcium, cholesterol, oral health and iron). The lessons consist of an introductory segment presented with online text and graphics. After reading this material, viewers have the option to complete one of four lesson activities. The activities provide opportunities for viewers to read further on the topic and are designed to reinforce key points of the lesson.
Arm/Group | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 371 | 373
Participants | 7 | 1

5. Secondary Outcome: Response to Survey Items Assessing Knowledge of the WIC Farmers' Market Nutrition Program Using a True/False Format.
Description: Index of Knowledge of the FMNP Score range: 0-6 Higher scores indicates greater knowledge
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 4.88 (.08) | 4.45 (.08) | 5.07 (.07) | 4.85 (.07)
  3-month follow-up | 4.79 (.09) | 4.71 (.09) | 5.07 (.08) | 5.01 (.08)
  6-month follow-up | 4.67 (.10) | 4.82 (.10) | 5.11 (.09) | 4.90 (.09)

6. Secondary Outcome: Response to an Item Assessing Knowledge of WIC-authorized Farmers' Markets Using a Yes/no Format.
Description: Knowledge of a farmers' market with farmers approved by WIC to accept WIC farmers' Market Nutrition Program and Cash Value vouchers Scores: No (0) and yes (1). Higher scores (yes responses) indicate that the respondent knows of a farmers' market with farmers approved by WIC to accept WIC farmers' Market Nutrition Program and Cash Value vouchers. Odds ratios and 95% confidence intervals indicate the likelihood of the outcome (knowledge of such markets) among those in the WIC Fresh Start (FMNP) arm relative to the comparator arm.
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Population: The WIC Fresh Start Program (FMNP) arm is being compared with each other study arm for this analysis.
Measure: Number (95% Confidence Interval); unit: Odds ratio
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 201
Odds ratio
  Posttest | 1.85 [.95 to 3.58] | 4.51 [2.42 to 8.42] | 2.44 [1.29 to 4.62]
  3-month follow-up | 2.25 [1.04 to 4.90] | 5.06 [2.40 to 10.69] | 2.18 [1.01 to 4.71]
  6-month follow-up | 1.50 [.64 to 3.52] | 4.41 [2.00 to 9.71] | 1.52 [.68 to 3.42]

7. Secondary Outcome: Response to Survey Items Assessing Attitudes Towards Farmers' Market Fruits and Vegetables Using 7-point Likert Rating Scales.
Description: Attitudes towards Farmers' Market Fruits and Vegetables Score range: 6-42 Higher scores indicate more favorable attitudes
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 12.27 (.66) | 10.70 (.65) | 11.05 (.59) | 11.10 (.60)
  3-month follow-up | 11.92 (.70) | 11.48 (.73) | 10.24 (.65) | 11.42 (.63)
  6-month follow-up | 12.03 (.78) | 11.45 (.81) | 10.19 (.73) | 12.27 (.70)

8. Secondary Outcome: Response to Survey Items Assessing Awareness of Locally Grown, Seasonal Fruits and Vegetables Using a Yes/no Format.
Description: Familiarity with Locally Grown Seasonal Items Score range: 0-3 Higher scores indicate greater familiarity
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 2.81 (.05) | 2.70 (.05) | 2.82 (.04) | 2.67 (.04)
  3-month follow-up | 2.79 (.05) | 2.76 (.05) | 2.86 (.05) | 2.75 (.05)
  6-month follow-up | 2.81 (.06) | 2.80 (.06) | 2.93 (.05) | 2.70 (.05)

9. Secondary Outcome: Response to Survey Items Assessing Fruit and Vegetable Food Safety Skills Using 7-point Likert Rating Scales.
Description: Fruit and Vegetable Food Safety Skills Score range: 19-85 Higher scores indicate greater skills
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 67.80 (.92) | 63.99 (.91) | 68.47 (.82) | 63.49 (.84)
  3-month follow-up | 66.70 (.98) | 64.13 (1.01) | 66.58 (.91) | 62.59 (.88)
  6-month follow-up | 69.11 (1.10) | 66.13 (1.13) | 66.44 (1.02) | 65.23 (.80)

10. Secondary Outcome: Response to Survey Items Assessing Farmers' Market Asking Skills Using a Yes/no Format.
Description: Farmers' Market Asking Skills Score range: 0-3 Higher scores indicate greater skills
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | .55 (.33) | .45 (.32) | .92 (.25) | 1.14 (.28)
  3-month follow-up | .49 (.35) | 1.31 (.56) | .85 (.33) | .68 (.34)
  6-month follow-up | 1.29 (.40) | 1.30 (.59) | 1.31 (.45) | 1.60 (.46)

11. Secondary Outcome: Response to Survey Items Assessing Positive Outcome Expectations for Consuming Locally Grown Fruits and Vegetables Using a Yes/no Format.
Description: Positive Outcome Expectations for Consuming Locally Grown Fruit and Vegetables Score range:0-3 Higher scores indicate more favorable ratings
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 2.91 (.03) | 2.86 (.03) | 2.93 (.03) | 2.88 (.03)
  3-month follow-up | 2.85 (.03) | 2.92 (.04) | 2.92 (.03) | 2.90 (.03)
  6-month follow-up | 2.95 (.04) | 2.97 (.04) | 2.97 (.04) | 2.96 (.03)

12. Secondary Outcome: Response to an Item Assessing Whether the Participant Ever Purchased Fruits and Vegetables at a Farmers' Market Using a Yes/no Format.
Description: Lifetime Farmers' Market Fruit and Vegetable Purchases Scores: No (0), Yes (1). Higher scores (yes responses) indicate indicate that the respondent has ever purchased fruits and vegetables at a farmers' market. Odds ratios and 95% confidence intervals indicate the likelihood of the outcome (having ever purchased fruits and vegetables at a farmers' market) among those in the WIC Fresh Start (FMNP) arm relative to the comparator arm.
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Population: The WIC Fresh Start (FMNP) arm is being compared with the three other study arms.
Measure: Number (95% Confidence Interval); unit: Odds ratio
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 201
Odds ratio
  Posttest | 1.78 [.90 to 3.53] | 1.06 [.52 to 2.17] | 1.31 [.66 to 2.58]
  3-month follow-up | 8.70 [3.06 to 25.00] | 6.04 [2.06 to 17.76] | 3.36 [1.13 to 10.04]
  6-month follow-up | 1.65 [.61 to 4.48] | 1.50 [.53 to 4.24] | 1.05 [.37 to 2.96]

13. Secondary Outcome: Response to Survey Items Assessing Farmers' Market Fruit and Vegetable Preparation Skills Using 7-point Likert Rating Scales.
Description: Farmers' Market Fruit and Vegetable Preparation Skills Score range:12-84 Higher scores indicate greater skills
Time Frame: 2 weeks
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 72.50 (.02) | 71.72 (.91) | 72.19 (.82) | 69.63 (.84)
  3-month follow-up | 73.06 (.98) | 72.53 (1.01) | 72.33 (.90) | 71.55 (.97)
  6-month follow-up | 73.27 (1.09) | 73.07 (1.13) | 72.99 (1.01) | 71.40 (.97)

14. Secondary Outcome: Response to an Item Assessing Whether the Participant Purchased Fruits and Vegetables at a Farmers' Market in the Past Two Weeks Using a Yes/no Format.
Description: Recent Farmers' Market Fruit and Vegetable Purchases Scores: No (0), Yes (1). Higher scores (yes responses) indicate that the respondent purchased fruits and vegetables at a farmers' market in the past two weeks. Odds ratios and 95% confidence intervals indicate the likelihood of the outcome (having purchased fruits and vegetables at a farmers' market in the past two weeks) among those in the WIC Fresh Start (FMNP) arm relative to the comparator arm.
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Population: The WIC Fresh Start (FMNP) arm is being compared with the three other study arms.
Measure: Number (95% Confidence Interval); unit: Odds ratio
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 201
Odds ratio
  Posttest | 1.07 [.59 to 1.96] | 2.18 [1.14 to 4.16] | 1.25 [.71 to 2.21]
  3-month follow-up | .81 [.39 to 1.69] | 2.23 [.91 to 5.47] | 1.07 [.53 to 2.16]
  6-month follow-up | .44 [.17 to 1.13] | .68 [.25 to 1.90] | .78 [.30 to 2.04]

15. Secondary Outcome: Response to an Item Assessing Behavioral Intentions to Purchase Fruits and Vegetables at a Farmers' Market in the Next Two Weeks Using a Yes/no Format.
Description: Intentions to Purchase Fruits and Vegetables at a Farmers' Market Scores: no (0), Yes (1). Higher scores (yes responses) indicate that the respondent intends to purchase fruits and vegetables at a farmers' market in the next two weeks. Odds ratios and 95% confidence intervals indicate the likelihood of the outcome (intending to purchase fruits and vegetables at a farmers' market in the next two weeks) among those in the WIC Fresh Start (FMNP) arm relative to the comparator arm.
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Population: The WIC Fresh Start Program (FMNP) arm is being compared with the three other study arms.
Measure: Number (95% Confidence Interval); unit: Odds ratio
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 201
Odds ratio
  Posttest | 2.92 [1.41 to 6.02] | 5.16 [2.57 to 10.35] | 2.02 [.97 to 4.22]
  3-month follow-up | 2.04 [1.10 to 3.80] | 2.35 [1.25 to 4.41] | .98 [.52 to 1.87]
  6-month follow-up | .97 [.54 to 1.77] | .96 [.52 to 1.78] | 1.09 [.62 to 1.92]

16. Secondary Outcome: Response to Survey Items Assessing Knowledge of Locally Grown Seasonal Fruits and Vegetables Found at Farmers' Markets in July Using a Yes/no Format.
Description: Knowledge of Locally Grown Seasonal Fruits and Vegetables found at Farmers' Markets in July Score range:0-9 Higher scores indicate greater knowledge
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 8.08 (.11) | 7.99 (.11) | 8.22 (.11) | 7.80 (.10)
  3-month follow-up | 8.14 (.12) | 7.85 (.12) | 7.91 (.11) | 7.95 (.11)
  6-month follow-up | 8.17 (.30) | 7.98 (.14) | 8.17 (.12) | 8.05 (.12)

17. Secondary Outcome: Response to Survey Items Assessing Food-specific Knowledge Using a True/False Format
Description: Food-specific Knowledge Score range: 2-13 Higher scores indicate greater knowledge
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 10.42 (.14) | 9.47 (.14) | 10.31 (.13) | 9.33 (.13)
  3-month follow-up | 9.76 (.15) | 9.40 (.16) | 10.11 (.14) | 9.31 (.14)
  6-month follow-up | 9.83 (.17) | 9.92 (.18) | 10.01 (.16) | 9.44 (.15)

18. Secondary Outcome: Response to Survey Items Assessing Knowledge of Area Farmers' Markets
Description: Farmers' Market-specific Knowledge Score range:0-2 Higher scores indicate greater knowledge
Time Frame: Pretest, posttest, and 3- and 6-month follow-up
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
Number analyzed (Participants) | 178 | 172 | 193 | 201
Units on a scale
  Posttest | 1.37 (.08) | 1.39 (.09) | 1.65 (.07) | 1.51 (.08)
  3-month follow-up | 1.42 (.09) | 1.51 (.10) | 1.75 (.08) | 1.63 (.08)
  6-month follow-up | 1.51 (.10) | 1.35 (.11) | 1.69 (.09) | 1.68 (.09)

ADVERSE EVENTS:
Time Frame: Adverse events were monitored through study completion, i.e., for 6.5 months after baseline (baseline [pretest], posttest [two weeks after pretest] and 3 and 6 months after the posttest [6.5 months total]).
Arm/Group | WIC Fresh Start Program | Existing Online Health Education | WIC Fresh Start Program (FMNP) | Existing Online Health Education (FMNP)
All-Cause Mortality (participants affected / at risk) | 0/178 | 0/172 | 0/193 | 0/201
Serious Adverse Events (participants affected / at risk) | 0/178 | 0/172 | 0/193 | 0/201
Other Adverse Events (participants affected / at risk) | 0/178 | 0/172 | 0/193 | 0/201

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No